CLINICAL TRIAL: NCT06889129
Title: Effect of Local Heat and Cold Application in the Management of Peripheral Neuropathy in Breast Cancer Patients Receiving Chemotherapy: A Randomized Controlled Trial
Brief Title: Heat and Cold Therapy for Chemotherapy-Induced Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Sabahat Coşkun, Associate Professor Dr., Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bilecik16
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Keywords: Chemotherapy-Induced Peripheral Neuropathy (CIPN); breast cancer; Heat-cold application; Non-pharmacological methods
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study population will consist of breast cancer patients receiving taxane-based chemotherapy at the Daytime Chemotherapy Unit of a training and research hospital who meet the inclusion criteria. The sample size calculation was performed for the study. Before conducting the power analysis, the effect size needed to be determined. In this study, the effect size was derived from a similar previous study. Considering a Type I error (α) = 0.05 and Power (1-β) = 0.90, the effect size (d) was selected as 0.35 based on a one-way analysis of variance (ANOVA). Using G*Power 3.1.9.7, the minimum required sample size was calculated as 108 participants. Based on these parameters, the expected minimum sample size is 36 patients per group, with a total of 108 participants. However, considering potential dropouts during the study, a total of 114 patients are planned to be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): standard protocol=Patients in this arm will receive standard care without any additional interventions related to heat or cold application.
- Intervention group (Experimental): Cold-Heat application + standard protocol
  Interventions: Other: Experimental- Heat application; Other: Experimental-Cold application

INTERVENTIONS:
Other: Experimental- Heat application — Heat application + standard protocol=Hot Application Protocol
  Hot application will start daily and continue until the completion of 4 weeks. The area will be checked for infection, scar tissue, inflammation, and incision before the application, and the procedure will be explained to the patient and their family.
  The first application will be performed on the day the patient comes for chemotherapy, ensuring privacy by exposing only the application area and positioning the patient appropriately.
  Patients will be asked to sit on a chair or couch with both feet immersed in a foot bath containing 5 liters of water, approximately 5 cm above their ankles, every night before bed for one month. The water temperature will be 40°C. The application will last for 30 minutes.
  Patients will be advised to avoid contact with cold water, as well as the consumption of cold food and beverages.
  Other Names: Heat application
  Arms: Intervention group
Other: Experimental-Cold application — Cold application + standard protocol=Cold application will start daily and continue until the completion of 4 weeks.
  The area will be checked for infection, scar tissue, inflammation, and incision before the application, and the procedure will be explained to the patient and their family.
  The first application will be performed on the day the patient comes for chemotherapy, ensuring privacy by exposing only the application area and positioning the patient appropriately.
  Patients will be asked to sit on a chair or couch with both feet immersed in a foot bath containing 5 liters of water, approximately 5 cm above their ankles, every night before bed for one month. The water temperature will be between 23-26°C. The application will be performed by the researcher on the day the patient comes for weekly chemotherapy treatment.
  Patients will be advised to avoid contact with hot water, as well as the consumption of hot food and beverages.
  Other Names: Cold application
  Arms: Intervention group

SUMMARY:
Cancer patients undergoing chemotherapy experience various side effects depending on the treatment protocol used. Chemotherapy-Induced Peripheral Neuropathy (CIPN) is a dose-limiting and quality-of-life-reducing complication caused by chemotherapeutic agents. The development of neuropathy not only restricts patients' physical functions but may also lead to dose reduction or even the discontinuation of chemotherapy.

Among chemotherapeutic agents, taxanes are among the most common causes of neuropathy. Docetaxel and paclitaxel, which belong to the taxane group, are widely used chemotherapeutics in the treatment of breast cancer. The degeneration, which manifests as numbness, tingling, and burning sensations in the fingers and toes, progresses from the distal to the proximal end of peripheral nerve axons.

Although several potential agents have been clinically tested to prevent CIPN, no pharmacological agent other than duloxetine, which has limited efficacy, has been proven effective. A review of the literature reveals that non-pharmacological methods used in the management of peripheral neuropathy include transcutaneous electrical nerve stimulation (TENS), massage, exercise, heat and cold application, relaxation techniques, acupuncture, and reflexology. Studies investigating the effectiveness of local water baths in the treatment of neuropathy have reported that this approach is effective in managing neuropathic symptoms.

This randomized controlled trial aims to evaluate the effects of local heat and cold application on neuropathic symptoms in breast cancer patients undergoing chemotherapy. Data will be collected using the Patient Information Form, Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT), and the Heat and Cold Application Patient Follow-up Form. Assessments will be conducted in both the intervention and control groups before the intervention and at the end of a 4-week period.

This study is designed as a randomized controlled trial to determine the effects of local heat and cold application on neuropathy in patients with chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
Breast cancer patients undergoing chemotherapy experience various side effects depending on the treatment protocol used. The most common side effects include neutropenia, anemia, peripheral neuropathy, nausea, vomiting, diarrhea, constipation, and fatigue. Chemotherapy-Induced Peripheral Neuropathy (CIPN) is a dose-limiting and quality-of-life-reducing complication caused by chemotherapeutic agents. CIPN can develop either during or after chemotherapy and not only restricts patients' physical functions but may also lead to dose reduction or even treatment discontinuation.

Among chemotherapeutic agents, taxanes are among the most common causes of neuropathy. Docetaxel and paclitaxel, which belong to the taxane group, are widely used chemotherapeutics in the treatment of breast cancer. The incidence of taxane-induced peripheral neuropathy varies between 61% and 92%. Although taxane-induced neuropathy primarily presents with sensory symptoms, it is a toxicity that can also affect motor and autonomic functions. The degeneration, which manifests as numbness, tingling, and burning sensations in the fingers and toes, progresses from the distal to the proximal end of peripheral nerve axons. Neuropathy in the upper extremities typically appears later.

The neurotoxicity of taxane-induced neuropathy is dose-dependent, and progression ceases once the drug treatment is completed. Emerging symptoms can be prevented by reducing the drug dose or increasing the interval between doses. However, these adjustments may significantly compromise cancer treatment outcomes. Although numerous potential agents have been clinically tested to prevent chemotherapy-induced peripheral neuropathy, no pharmacological agent other than duloxetine, which has limited efficacy, has been proven effective.

A review of the literature reveals that non-pharmacological methods used in the management of peripheral neuropathy include transcutaneous electrical nerve stimulation (TENS), massage, exercise, heat and cold application, relaxation techniques, acupuncture, and reflexology. Medical baths have been used in the treatment of inflammatory and non-inflammatory rheumatic diseases, fibromyalgia, and chronic back pain, as well as for reducing fatigue and improving sleep regulation. In particular, foot bath studies have reported that foot baths increase blood circulation through vasodilation in peripheral blood vessels, improve sensory symptoms, stimulate the sense of touch, reduce sympathetic nerve activity, enhance skin permeability, promote microcirculation in cells, and support drug therapy.

A review of the literature indicates that very few studies have investigated the effects of foot baths on the management of peripheral neuropathy in cancer patients. Studies examining the effectiveness of local water baths in the treatment of neuropathy have reported that this approach is an effective strategy for managing neuropathic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Women with stage III-IV breast cancer receiving 4-7 cycles of taxane-based chemotherapy,
* Patients with chemotherapy-induced neuropathy symptoms,
* Residents of Ankara,
* Over 18 years older,
* No history of nerve damage or psychiatric illness,
* No central nervous system metastasis or disease,
* No irritation or ulceration in the skin area where the application will be made,
* No history of deep vein thrombosis,
* Not using anticoagulant medication,
* Able to speak, understand, and read/write in Turkish,
* Patients who consent to participate in the study will be included.

Exclusion Criteria

* Patients with a history of nerve damage or psychiatric illness,
* Ulcers or irritation in the area where the application will be made,
* Patients with peripheral neuropathy developed due to reasons other than chemotherapy,
* Patients who do not consent to participate in the study will be excluded.

Exclusion Criteria During the Study

* Patients whose taxane treatment protocol is changed,
* Patients who have less than four applications per week will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
1. Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) | At baseline (first visit) and at 4 weeks
  The Turkish validity and reliability of the scale were tested in breast cancer patients receiving taxane chemotherapy (n=430). The first section assesses sensory and motor symptoms (numbness, itching, burning, discomfort, cold sensitivity, pain, weakness, balance problems), with responses scored from 0 to 10. Higher scores indicate greater discomfort. In the second section, difficulties in daily activities (e.g., dressing, walking, working, exercising) are also rated from 0 to 10. The scale's overall Cronbach alpha is 0.87, with test-retest reliability ranging from 0.90 to 0.96. These results confirm that the scale is valid and reliable for the Turkish population.
Local Heat and Cold Application Patient Follow-up Form | At baseline (first visit) and at 4 weeks
  This form is designed to assess patients' adherence to local heat or cold application. During the heat or cold application process, patients will be followed up by phone to enhance their adherence to the program and ensure compliance. In addition, when patients come to receive their weekly chemotherapy doses, the application will be performed by the researcher.
  Patients will mark their heat or cold application status on the form while performing the application at home. The forms will be reviewed by the researcher when patients visit the hospital for chemotherapy treatment. Patients who perform the application less than four times per week will not be included in the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: SABAHAT COŞKUN, Doç.Dr., Study Director — Bilecik Şeyh Edebali Üniversity
Locations (1):
- Gulhane Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request, in accordance with ethical guidelines and with participant consent.
Supporting Information: Study Protocol, SAP